CLINICAL TRIAL: NCT02987062
Title: CRAFT - Multicenter Experience in Atrial Fibrillation Patients Treated With OAC (CRAFT)
Brief Title: MultiCenter expeRience in AFib Patients Treated With OAC (CRAFT)
Acronym: CRAFT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marcin Grabowski, Clinical Professor, Marcin Grabowski, Medical University of Warsaw, Medical University of Warsaw
Other Study IDs: CRAFT
Record Dates: First submitted 2016-11-30; First posted 2016-12-08 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Non-vitamin K Oral Anticoagulants; Vitamin K Antagonists; ROCKET-AF; RE-LY; ARISTOTLE
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Acenocoumarol: Patients with AF treated with acenocoumarol.
- Warfarin: Patients with AF treated with warfarin.
- Apixaban: Patients with AF treated with apixaban.
- Dabigatran: Patients with AF treated with dabigatran.
- Rivaroxaban: Patients with AF treated with rivaroxaban.

SUMMARY:
According to current guidelines for non-valvular atrial fibrillation treatment, the first line drugs are non-vitamin K oral anticoagulants (NOACs), which are preferred over vitamin K antagonists (VKAs). However, it is not clearly confirmed, how the success of NOACs approval trials (ROCKET-AF (rivaroxaban), RE-LY (dabigatran) and ARISTOTLE (apixaban) reflects on real-life clinical practice.

The aim of this study is to assess treatment of AF patients with oral anticoagulants (OACs) in an academic and district hospital, with regard to inclusion/exclusion criteria used in the clinical trials.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common arrhythmia associated with increased cardiovascular morbidity and mortality. An integral element of management of patients with AF is anticoagulation to prevent thromboembolic events. Non-vitamin K oral anticoagulants and vitamin K antagonists are two main drugs groups used in treatment.

Primary objective of the study is to assess the treatment of AF patients with OACs (the frequency of prescription of VKAs vs NOACs), compare the clinical characteristics of the real-life AF patients with populations included in the randomized clinical trials (ROCKET-AF, RE-LY and ARISTOTLE) and population gathered from the university department and the district hospital. Secondary objective of the study is to assess the long-term outcomes of patients with AF treated with OACs.

The CRAFT (MultiCenter expeRience in AFib patients Treated with OAC) is a multicenter retrospective analysis of hospital records of patients with AF managed in the First Department of Cardiology of Medical University of Warsaw and in John Paul II Western Hospital in Grodzisk Mazowiecki. Gathered data will include demographics, type of AF (valvular and non-valvular, as well as paroxysmal, persistent and permanent), medical history, baseline characteristics (i.e. blood pressure), laboratory investigations (blood tests, including renal and hepatic function), echocardiographic parameters and concomitant medications. Data will be collected from the moment of patient's discharge.

Each patient will be evaluated regarding to common and new scales assessing risk of thromboembolic (CHA2DS2-VASc ) and bleeding (HAS-BLED, HEMORR2HAGES, modifiable and non-modifiable risk factors for bleeding in anticoagulated patients basing on the current guidelines for AF treatment) events, as well as SAMeTT2R2 score to predict the quality of treatment on OACs.

ELIGIBILITY:
Inclusion criteria:

* paroxysmal, persistent, long-standing persistent or permanent AF
* valvular or non-valvular AF
* treatment with OACs (apixaban, dabigatran, rivaroxaban, acenocoumarol, warfarin)

Exclusion criteria:

* lack of OAC at hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with AF treated with VKAs (acenocoumarol, warfarin) and NOACs (apixaban, dabigatran, riwaroxaban), hospitalized in 2011-2016 years in the First Department of Cardiology of Medical University of Warsaw and hospitalized in 2014-2016 in the John Paul II Western Hospital in Grodzisk Mazowiecki, Poland.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of clinical characteristics of the real-life AF patients with populations included in the randomized clinical trials (ROCKET-AF, RE-LY and ARISTOTLE) | Through the study completion, an average of 3 months.
  Compared data will include: demographics, type of AF (valvular and non-valvular, as well as paroxysmal, persistent and permanent), medical history, baseline characteristics, laboratory investigations, echocardiographic parameters and concomitant medications. Each patient will be evaluated regarding to the modifiable and non-modifiable risk factors for bleeding basing on the current guidelines for AF treatment, CHA2DS2-VASc, HAS-BLED, HEMORR2HAGES scales and SAMeTT2R2 score.
Comparison of clinical characteristics of the AF patients treated in university department with population gathered from the district hospital | Through the study completion, an average of 3 months.
  Compared data will include: demographics, type of AF (valvular and non-valvular, as well as paroxysmal, persistent and permanent), medical history, baseline characteristics, laboratory investigations, echocardiographic parameters and concomitant medications. Each patient will be evaluated regarding to the modifiable and non-modifiable risk factors for bleeding basing on the current guidelines for AF treatment, CHA2DS2-VASc, HAS-BLED, HEMORR2HAGES scales and SAMeTT2R2 score.

SECONDARY OUTCOMES:
Assessment of the frequency of VKAs vs NOACs prescription in AF patients treatment of with OACs | Through the study completion, an average of 3 months.
Assessment of long-term outcomes (death, hospitalizations, minor/major/life-threatening bleeding, thromboembolic events) | Through the study completion, an average of 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Opolski, Professor, Study Chair — 1st Department of Cardiology Medical University of Warsaw; Marcin Grabowski, PhD, Study Chair — 1st Department of Cardiology Medical University of Warsaw
Locations (2):
- Poland (2):
  - 1st Department of Cardiology Medical University of Warsaw, Warsaw, Mazowiecki
  - John Paul II Western Hospital, Grodzisk Mazowiecki

REFERENCES:
- [Derived] Maciejewski C, Ozieranski K, Basza M, Barwiolek A, Ciurla M, Bozym A, Krajsman MJ, Lodzinski P, Opolski G, Grabowski M, Cacko A, Balsam P. Practical use case of natural language processing for observational clinical research data retrieval from electronic health records: AssistMED project. Pol Arch Intern Med. 2024 May 28;134(5):16704. doi: 10.20452/pamw.16704. Epub 2024 Mar 19. PMID 38501989
- [Derived] Balsam P, Tyminska A, Ozieranski K, Zaleska M, Zukowska K, Szepietowska K, Maciejewski K, Peller M, Grabowski M, Lodzinski P, Koltowski L, Praska-Oginska A, Zaboyska I, Bednarski J, Filipiak KJ, Opolski G. Randomized controlled clinical trials versus real-life atrial fibrillation patients treated with oral anticoagulants. Do we treat the same patients? Cardiol J. 2020;27(5):590-599. doi: 10.5603/CJ.a2018.0135. Epub 2018 Nov 8. PMID 30406937